CLINICAL TRIAL: NCT03663816
Title: Villency - Proof of Action: Foot Device, Balance and Sway, Kinematics of Walking
Brief Title: Villency-Proof of Action: Foot Device, Balance and Sway, Kinematics of Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Villency Design Group, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCR18420; AGR00011966 (Other: University of Florida)
Record Dates: First submitted 2018-08-24; First posted 2018-09-10 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Balance
Keywords: shoe insert; orthotics; sway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy men and women (Experimental): Participants will serve as their own control. Balance and gait measures will be collected during an initial visit and after one week of using the experimental foot device
  Interventions: Device: experimental foot device

INTERVENTIONS:
Device: experimental foot device — Appropriately-designed, stimulatory - but not mechanically supportive -device to enhance control of balance, postural sway and key features of walking gait in healthy people.
  Other Names: proprioceptive foot device

SUMMARY:
This study involves the use of a newly designed shoe insole device (also referred to as a foot insole device) similar to various shoe insoles or inserts you can buy at a store or pharmacy.

DETAILED DESCRIPTION:
This study involves the use of a newly designed shoe insole device (also referred to as a foot insole device) similar to various shoe insoles or inserts you can buy at a store or pharmacy. Healthy participants will wear this insole device in their own athletic/tennis shoes over the course of one week. There are two key purposes of this study: 1. To determine how using this insole device for 1 week may effect a healthy individual's balance and postural sway while standing; and 2. To determine how using this insole device for 1 week may effect how an individual walks (gait), how hard they hit the ground as they walk, and foot pressure patterns with each step. Each individual's balance, postural sway, and walking gait (how you walk) will be analyzed before and after wearing the shoe insole device for the one-week time period.

ELIGIBILITY:
Inclusion Criteria:

● Willing to maintain current level of physical activity during the study period of a week (no increase or decrease of activity level).

Exclusion Criteria:

* Moderate or severe obesity (body mass index >35kg/m2)
* Known diagnosis of cardiovascular, orthopaedic, or neurological conditions, uncontrolled diabetes, or any condition that impacts normal walking ability
* Any current ankle, knee, hip or low back pain
* Currently using any knee or ankle brace on a regular basis for joint pains
* Severe back pain, prior spinal fusion or spinal deformity that would affect gait
* Major cardiac or pulmonary conditions and any orthopedic limitation that precludes their ability to independently walk for 10 minutes or longer
* Any major orthopedic injury within the prior 12 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Vincent, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Men and Women
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Men and Women
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — All races accepted
  Participants
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 11
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Center of Mass Displacement (Sway) During Standing
Description: Two-foot stance, Single foot balance, and Tandem stance- Once the data are collected, calculations of center of mass displacement (in cm) will be determined. These values will provide insight about direction of sway and how quickly sway occurs during these three balance conditions.
Time Frame: At 1 week of acclimation
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Healthy Men and Women
Number analyzed (Participants) | 15
centimeters | .62 (.24)

2. Primary Outcome: Center of Variability Displacement During Standing
Description: Two-foot stance, Single foot balance, and Tandem stance- the variability of displacement and area (cm2) will be determined
Time Frame: At 1 week of acclimation
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Healthy Men and Women
Number analyzed (Participants) | 15
centimeters | .75 (.13)

3. Primary Outcome: Center of Peak Speed of Displacement.
Description: Two-foot stance, Single foot balance, and Tandem stance- and the peak speed of displacement (cm per second) will be determined.
Time Frame: At 1 week of acclimation
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Healthy Men and Women
Number analyzed (Participants) | 15
centimeters per second | 8.58 (3.63)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Healthy Men and Women
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03663816/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03663816/ICF_000.pdf